CLINICAL TRIAL: NCT03929939
Title: Neural Control and Cardiac-Vascular Function in Women With PTSD (VA Psychological Assessment)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Collaborators: University of Texas Southwestern Medical Center (Other); Texas Health Resources (Other)
Responsible Party: Principal Investigator, Geetha Shivakumar, Principal Investigator, North Texas Veterans Healthcare System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-061
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Exercise; Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Modification Group (Experimental)
  Interventions: Behavioral: Exercise training and healthy eating (overseen by IEEM research team)
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Exercise training and healthy eating (overseen by IEEM research team) — Exercise Training: A "personalized" training program will be developed for participants. Based on maximal steady state heart rate and resting heart rate, three training zones (recovery, base pace, and maximal steady state) will be determined. The target heart rate for each training zone will be set for each patient. The majority of training sessions during the early phase of the program will be prescribed as "base pace" with target heart rate equivalent to about 75% of maximal. Initially, patients will train 3 times per week for 20-30 minutes per session by walking, jogging or swimming. As the patients become relatively fit, the duration of the base training sessions will be prolonged, and subsequently sessions of increased intensity (i.e., maximal steady state) will be added.
  Healthy Eating: Participants will be provided with dietary advice consistent with the American Heart Association guidelines (D.A.S.H. diet eating plan).
  Arms: Lifestyle Modification Group

SUMMARY:
The purpose of this research is 1) to investigate the role of the sympathetic nervous system and cardiac-vascular function in women with PTSD; and 2) to determine whether lifestyle modifications (exercise training and healthy eating) would be effective in reducing sympathetic activity, improving cardiovascular function, and improving psychiatric and quality of life outcomes in women with PTSD. It is hypothesized that (1) women with PTSD will have over-activation of the sympathetic nervous system and impaired cardiac-vascular function compared with women who are trauma free, and (2) lifestyle modifications can reduce sympathetic activity, improve cardiac-vascular function, and improve psychiatric symptoms and quality of life in women with PTSD.

DETAILED DESCRIPTION:
This is a collaborative study between the Institute for Exercise and Environmental Medicine (IEEM; Texas Health Resources/University of Texas Southwestern medical Center) and VA North Texas Healthcare System (VANTHCS). The overall study was conceptualized and initiated by Dr. Qi Fu and her research team at the IEEM. IEEM researchers will be responsible for recruitment of non-veteran women without a diagnosis of PTSD, physiological assessments, and the lifestyle modification intervention. VANTHCS researchers will be responsible for recruitment of women veterans with PTSD and psychological assessments. The procedures taking place at VANTHCS (recruitment of women Veterans with PTSD and psychological assessments) will fall under a separate study (overseen by VANTCHS IRB and RDC) and will not include the procedures and intervention that will take place at the IEEM (which will be overseen by a separate IRB). Data will be shared between the sites per data sharing agreement. This clinical trials entry reflects the VANTHCS study. Outcome measures gathered by the IEEM research team are included in this entry due to the data sharing agreement.

ELIGIBILITY:
Inclusion Criteria:

1. Be either a female veteran with a current diagnosis of PTSD (for the PTSD group) or a female non-veteran without a current diagnosis of PTSD (for the non-PTSD control group).
2. Be between the ages of 18-65.
3. Sedentary (exercises less than three times a week for thirty minutes or less).

Exclusion Criteria:

1. Any evidence of cardiopulmonary and neurological diseases by history or by physical examination.
2. Chronic kidney disease (serum creatinine > 1.5 mg/dL).
3. Peripheral vascular disease.
4. Peripheral neuropathy.
5. Current substance use disorder other than tobacco related.
6. Endurance-trained athletes due to the effects of exercise training on sympathetic neural control and cardiac-vascular function.
7. Current pregnancy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Muscle Sympathetic Nerve Activity (MSNA; Data collected by IEEM) | +PTSD vs. -PTSD baseline comparison; Changes from baseline following 12-week intervention
  Muscle sympathetic nerve activity will be measured using microneurography at the peroneal nerve.
Clinician Administered Posttraumatic Stress Disorder Scale - 5 (CAPS-5; Data collected by VANTHCS) | Changes from baseline following 12-week intervention
  CAPS-5 is a 30-item structured interview that corresponds to the DSM-5 diagnosis for PTSD. The instrument is used to make a current or lifetime diagnosis of PTSD, as well as assess symptom severity. Total symptom severity scores range from 0 to 80. A higher score indicates greater symptom severity. Individual symptom severity scores range from 0 (absent) to 4 (extreme/incapacitating) and are based on symptom frequency and intensity.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5; Data collected by VANTHCS) | Changes from baseline through 12-week intervention
  Self-report measure of PTSD symptoms
Quick Inventory for Depressive Symptomatology-self report (QIDS- SR16; Data collected by VANTHCS) | Changes from baseline through 12-week intervention
  Self-report measure of depression symptom severity. Total scores range from 0-27. A higher score indicates greater symptom severity.
Concise Health Risk Tracking Scale - self-report module (CHRT; data collected by VANTHCS) | Changes from baseline through 12-week intervention
  The CHRT-SR is a 16-item self-report measure that assesses suicidal propensity and risk. All items are scored on a 5-point Likert scale ranging from "strongly disagree" (0) to "strongly agree" (4). The propensity score (items 1-13) assesses pessimism, helplessness, perceived lack of social support, and despair. The propensity score may range from 0 to 52, with higher scores showing higher levels of suicidal propensity. The risk score (items 14-16) assess thoughts and plans of killing oneself. The risk score may range from 0-12, with a higher score showing higher levels of suicidal thoughts.
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF; data collected by VANTHCS) | Changes from baseline through 12-week intervention
  The Q-LES-Q-SF is a 16 item self-report measure that assesses perceived quality of life. All items are scored on a 5-point Likert scale ranging from "very poor" (1) to "very good" (5). raw total score is created by summing the first 14 items. The last two items are standalone items and not included in the total score. Raw total score ranges from 14-70. The raw total score is transformed into a percentage maximum possible score using the following formula: (raw total score - minimum score)/(maximum possible raw score-minimum score). Percentage maximum ranges from 0% to 100, with a lower percentage indicating worse perceived quality of life.
36-Item Short Form Health Survey (SF-36; Data collected by IEEM) | +PTSD vs. -PTSD baseline comparison; Changes from baseline following 12-week intervention
  The SF-36 is a 36-item self-report measure of general health status. The measure includes multi-item scales to measure the following 8 dimensions: physical functioning; role limitations due to physical health problems; bodily pain; social functioning; general mental health; role limitations due to emotional problems; vitality, energy, or fatigue; and general health perceptions. All items are scored so that a higher score indicates a more favorable health state. The SF-36 produces two sets of scores: a profile of eight sections scores, and two summary scores (physical component scores [PCS] and mental component scores [MCS].
Endothelial function (data collected by IEEM) | +PTSD vs. -PTSD baseline comparison; Changes from baseline following 12-week intervention
  Measured using flow-mediated vasodilation
Arterial stiffness (Data collected by IEEM) | +PTSD vs. -PTSD baseline comparison; Changes from baseline following 12-week intervention
  Central and peripheral pulse wave velocity measured using arterial tonometry
Systolic and diastolic cardiac function (Data collected by IEEM) | +PTSD vs. -PTSD baseline comparison; Changes from baseline following 12-week intervention
  Measured using echocardiogram
Physical Fitness (Data collected by IEEM) | Changes from baseline following 12-week intervention
  Peak oxygen uptake (Douglas bag method) during submaximal and maximal treadmill test

CONTACTS AND LOCATIONS:
Overall Officials: Geetha Shivakumar, MD, MS, Principal Investigator — Dallas VA Medical Center
Locations (2):
- United States (2):
  - Dallas VA Medical Center, Dallas, Texas
  - The Institute for Exercise and Environmental Medicine, Dallas, Texas

DOCUMENTS (1):
  • Informed Consent Form (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT03929939/ICF_000.pdf